CLINICAL TRIAL: NCT06860139
Title: Developing a Health Literacy Intervention for Immigrant Kidney Transplant Recipients
Acronym: IMMIHEALTH
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse Sor-Ost (Helse Sør-Øst) (Unknown)
Responsible Party: Principal Investigator, Kari Gire Dahl, Doctor, Oslo University Hospital
Other Study IDs: 23/01097; 2023027 (Other: Helse Sor-Ost (Helse Sør-Øst))
Record Dates: First submitted 2025-02-04; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Transplant Recipient (Kidney)
Keywords: Health literacy intervention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Two different groups of patients and two groups of nurses are included.: Before intervention development:
  * Thirteen patients are interviewed three times following the kidney transplantation (during the first week, before transfer to the local hospital, about 4-6 weeks following kidney transplantation, and after 3 to 6 months). Nurses in three wards that follow these patients are interviews in five focus groups.
  * The intervention will then be developed in co-creation with nurses and patients.
  Optimizing intervention:
  - In the optimizing process, the interviews and focus group interviews are repeated to explore satisfaction and assess the need for change.
  Interventions: Behavioral: Health literacy intervention

INTERVENTIONS:
Behavioral: Health literacy intervention — The intervention will be developed in co-creation with patients and nurses in the clinic, based on their needs.

SUMMARY:
The goal of this complex interventions study is to improve health literacy (HL), medication adherence and patient education outcomes in immigrant kidney transplant recipients (KTRs). Furthermore, we aim to strengthen HL sensitivity and cultural competence in nurses providing patient education. The main questions we aims to answer are:

1. What are immigrant KTRs HL strengths and needs, medication adherence and outcomes after patient education in three important transitions following kidney transplantation: the first postoperative phase (3-7 days post-transplantation), preparing for transfer to local hospital (6-8 weeks post-transplantation), and adapting to the home context (3-6 months post-transplantation).
2. What experiences, competence and competence needs does the nurses that engage in patient education to immigrant KTRs post-transplant have?
3. Will a tailored intervention increase HL, medication adherence, and outcomes after patient education in immigrant KTXs and organizational HL and cultural competence in nurses?

Qualitative methods will be used to develop and optimize the intervention.

* Patients will be invited to three individual interviews in the three postoperative phases.
* Nurses in three wards (surgery, medical and outpatient ward) are asked to participants in focus group interviews.
* The interviews will be used to define needs and build the intervention. Ideas to the intervention will be discussed in workshops with nurses, the project group and user participants.
* Parts of the intervention will be tested in the clinic followed by 'think aloud interviews' where both the nurse and the patient are asked to speak freely about their experiences using the intervention.
* The intervention will be evaluated by repeating the interviews with patient and focus group interviews with nurses.
* The intervention will be feasibility tested.

ELIGIBILITY:
Inclusion Criteria:

* Immigrant kidney transplant recipients in Norway. Immigrant defined as a person that has immigrated to Norway and that has two parents and two grandparents born in another country than Norway.

Exclusion Criteria:

* Patients from high-income countries, as defined by the Global Burden of Disease (GBD) framework. The GBD study is the largest and most comprehensive effort to quantify health loss across places and over time (https://www.healthdata.org/research-analysis/gbd). High income countries are western Europe, North America, Australia, New Zealand, Japan, Brunei, Republic of Korea, and Singapore (https://ghdx.healthdata.org/countries). National and international studies report that people with background from low-income countries have lower sociodemographic scores and lower health literacy levels. Therefore, the study will focus on these patients. The majority of immigrant kidney transplant recipients in Norway are from low-income countries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Immigrant kidney transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
All outcomes are defined from qualitative data (Individual patient interviews and focus group interviews with nurses). | November 2027
  Patients experiences from patient education, health literacy (strengths, challenges, expectations and needs), information about medication adherence and transplant knowledge will be collected using qualitative interviews. The interview guide is developed using the conversational health literacy tool (CHAT), that involve questions about health literacy. The tool is flexible and adaptable to the transplant context and will also involve questions regarding medication adherence and transplant knowledge.
  Nurses experience from giving patient education will be collected through focus group interviews. The interview guide involves the following four main themes: experiences giving patient education to immigrant kidney transplant recipient, giving patient education using an interpreter, competence and competence needs and documenting patient education with immigrant patients.
  Quantitative measures are not used.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No